CLINICAL TRIAL: NCT01695161
Title: Corneal-Compensated Intraocular Pressure, Corneal Hysteresis and Corneal Resistance Factor Measurements Performed With the Ocular Response Analyzer and Their Correlation to Conventional Goldmann Applanation Tonometry.
Brief Title: Non-invasive Assessment of Intraocular Pressure in MPS by Use of the Ocular Response Analyzer.
Acronym: MPSORA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Johannes Gutenberg University Mainz (Other)
Responsible Party: Principal Investigator, Susanne Pitz, MD, Johannes Gutenberg University Mainz
Other Study IDs: MZ-MPS-2012-01
Record Dates: First submitted 2012-09-25; First posted 2012-09-27 (Estimated); Last update posted 2013-03-01 (Estimated); Status verified 2013-02

CONDITIONS: Mucopolysaccharidosis; Fabry Disease
Keywords: Mucopolysaccharidosis; Fabry disease
MeSH Terms: conditions — Mucopolysaccharidoses; Fabry Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- mucopolysaccharidosis: mucopolysaccharidosis
- Fabry disease: Fabry disease
- healthy controls: healthy controls

SUMMARY:
The aim of the present study is to compare intraocular pressure (IOP) values assessed with Ocular Response Analyzer to the classical gold standard of IOP measurement, to Goldmann applanation tonometry by mucopolysacchyridosis-, Fabry-patients and healthy controls. We want to investigate biomechanical characteristics of the cornea and their influence on the IOP-measurements.

ELIGIBILITY:
Inclusion Criteria:

* MPS I, II, IV, VI patients with at least grade 3 of corneal clouding (Couprie et al.)
* Fabry patients with cornea verticillata > grade 1
* Age ≥ 12 years
* Patient is able to comply with the study procedure
* Patient has consented to be in the trial
* Ability to fixate a target

Exclusion Criteria:

* History of corneal transplantation or refractive surgery
* Corneal pathologies other than MPS-associated corneal opacity
* Corneal, conjunctival or intraocular inflammation

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: 25 eyes of MPS patients 25 eyes of Fabry patients 25 eyes of healthy age matched controls (a difference of ± 5 years in the mean between both groups is accepted)
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2012-09; Primary Completion 2013-09 (Estimated)

PRIMARY OUTCOMES:
agreement between ccIOP and GAT in MPS, Fabry and healthy controls | Sep 2013 (anticipated)
  Evaluation of agreement between ccIOP and GAT in MPS, Fabry and healthy controls

CONTACTS AND LOCATIONS:
Overall Officials: Susanne Pitz, MD, Principal Investigator — Department of Ophthalmology, University Medical Center, Johannes Gutenberg-
Locations (1):
- Department of Ophthalmology, University Medical Center, Johannes Gutenberg-, Mainz, Germany

REFERENCES:
- [Derived] Wasielica-Poslednik J, Politino G, Schmidtmann I, Lorenz K, Bell K, Pfeiffer N, Pitz S. Influence of Corneal Opacity on Intraocular Pressure Assessment in Patients with Lysosomal Storage Diseases. PLoS One. 2017 Jan 12;12(1):e0168698. doi: 10.1371/journal.pone.0168698. eCollection 2017. PMID 28081172